CLINICAL TRIAL: NCT07376746
Title: Improving ADHD Core Symptoms and Individual Quality of Life With Dietary APproaches Through Microbiota-Gut-Brain Signalling
Brief Title: Improving ADHD Symptoms and Quality of Life Through Diet
Acronym: ADAPT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College Cork (Other)
Collaborators: APC Microbiome Ireland, UCC (Other)
Responsible Party: Principal Investigator, John Cryan, PhD, University College Cork
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: APC199
Record Dates: First submitted 2026-01-21; First posted 2026-01-29 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: ADHD
Keywords: Psychobiotic diet; ADHD; Fermented foods; Gut-Brain Axis; Dietary fibre
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: This is a double-blind study where both participants and outcomes assessors are blinded to group allocation. Randomization and assignment to dietary groups will be conducted by a staff member not involved in study visits or data analysis as well as the organisation of fermented food deliveries. Dietary counselling will be delivered by a separate dietitian who is aware of group allocation but has no role in outcome assessment or other study procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- No ADHD/Combined Diet (Experimental): Participants without ADHD will receive a combined diet (fermented foods and high fiber)
  Interventions: Other: Combined diet
- No ADHD/Control diet (No Intervention): Participants without ADHD will receive dietary education based on the healthy eating guidelines provided by the Health Service Executive (HSE).
- ADHD/Control diet (No Intervention): Participants with ADHD will receive dietary education based on the healthy eating guidelines provided by the Health Service Executive (HSE).
- ADHD/Combined diet (Experimental): Participants with ADHD will receive a combined diet (fermented foods and high fiber)
  Interventions: Other: Combined diet

INTERVENTIONS:
Other: Combined diet — Participants will receive dietary education to increase their fibre intake to 25-30g/day and include 3 to 4 portions of fermented foods to their normal diet.
  Arms: ADHD/Combined diet; No ADHD/Combined Diet

SUMMARY:
The goal of this randomised controlled trial is to evaluate whether a specific dietary intervention can reduce core symptoms of Attention-Deficit/Hyperactivity Disorder (ADHD) in adults aged 18 to 50 years. The study also aims to understand how changes in diet may influence quality of life, neurocognitive function, and gut-brain signaling through the microbiota.

The main questions it aims to answer are:

1. Does a high-fiber, fermented food-based diet reduce ADHD core symptoms over a 12-week period, as measured by the Conners' Adult ADHD Rating Scale (CAARS)?
2. Does the diet improve neurocognitive function, mood, food reward, individual goals, and other quality-of-life outcomes?
3. How does the diet affect gut microbial composition, inflammation, and stress-related biomarkers?
4. Is the diet well-accepted and feasible to follow?

Researchers will compare a combination intervention diet (high in fiber and fermented foods) to a control diet based on general healthy eating guidelines to assess differences in symptom improvement and biological outcomes.

Participants will:

1. Complete six study visits over a 24-week period (screening, baseline, weeks 4, 8, 12, and optional follow-up at week 24).
2. Be randomly assigned to one of two dietary groups after baseline assessments.
3. Provide stool, saliva, urine, and blood samples at multiple timepoints.
4. Undergo cognitive testing and EEG recording to assess brain function.
5. Wear a wristband to track sleep and activity patterns.
6. Use a nutrition app to log dietary intake and receive weekly dietary support.
7. Complete validated questionnaires on ADHD symptoms, mood, eating behavior, gastrointestinal health, sleep, and lifestyle factors. Feasibility and acceptability of following the diet will also be self-reported.

This study includes both adults diagnosed with ADHD and matched controls without a psychiatric condition to better understand the mechanisms and potential differential responses to dietary intervention.

DETAILED DESCRIPTION:
This is a participant-blind, observer-blind, randomized, controlled, parallel-group trial designed to evaluate the effects of a dietary intervention on core symptoms of Attention-Deficit/Hyperactivity Disorder (ADHD) and related neurocognitive and physiological parameters in adults. The study also investigates the mechanisms underlying these effects, with a focus on the microbiota-gut-brain axis.

A total of 200 participants (100 adults with a diagnosis of ADHD/ADD and 100 healthy controls) aged 18 to 50 years will be recruited and randomized to one of two dietary arms:

1. A combination intervention diet rich in fiber and fermented foods.
2. A control diet based on general healthy eating guidelines following the Irish Food Pyramid.

The intervention period lasts for 12 weeks, followed by a 12-week optional follow-up.

The primary objective is to assess the change in ADHD symptoms, measured using the Conners' Adult ADHD Rating Scale (CAARS), from baseline to week 12. Secondary outcomes include changes in cognition, mood, quality of life, and individual goal attainment. Tertiary outcomes include alterations in eating behavior, sleep, activity patterns, diet feasibility and acceptability, gut microbiota composition and diversity, microbial metabolites (e.g., short-chain fatty acids), systemic inflammatory markers, and stress biomarkers (cortisol).

Study Design and Procedures

Participants will complete six study visits:

Visit 1 (Screening): Consent, eligibility assessment via structured psychiatric interview (MINI and DIVA for ADHD; MINI and ASRS for controls as well as assessing other in- and exclusion criteria), baseline sociodemographic and health data, dietary logging app setup, and instructions for pre-visit biological sample collection (stool, urine, saliva).

Visit 2 (Baseline, pre-intervention): Biological sample collection, cognitive testing, EEG (resting-state, response inhibition, and food cue responsivity), anthropometry, blood pressure, and detailed questionnaires on ADHD symptoms, mood, cognition, sleep, lifestyle, and individual goal setting. Participants are randomized and receive individualized dietary advice and guidance based on their group assignment.

Visits 3 and 4 (Week 4 and Week 8): Collection of biological samples, lifestyle and symptom questionnaires, adherence reinforcement with the dietitian, and adverse event monitoring. Body weight, circumferences, and blood pressure are reassessed.

Visit 5 (Week 12, post-intervention): Full reassessment mirroring Visit 2. Participants are debriefed, compensated, and provided with post-intervention materials. Perceived allocation (control vs. intervention) and acceptability/feasibility of the diet are also evaluated.

Visit 6 (Optional follow-up at Week 24): Evaluation of sustained effects on ADHD symptoms, quality of life, adherence, and feasibility. Stool sample is collected, anthropometry is repeated, and diet is logged again.

During the intervention, participants track their diet using a smartphone app (Nutritics/Libro) and receive weekly email support. Participants also receive personalized dietary advice according to their group allocation: a minimum of 25 grams of fiber and 3 servings of fermented foods per day for those in the combined diet group; or, for those in the control diet group, adherence to the standard food pyramid (daily portions include 5-7 servings of fruits and vegetables, 3-5 servings of whole grains, 2 servings of lean protein such as meat, fish, eggs, or legumes, 3 servings of low-fat dairy, and limited intake of fats, oils, and sweets).

Biological samples (stool, saliva, urine, blood) will be collected at multiple timepoints. Stool samples will be used for microbiota profiling (16S rRNA sequencing and metagenomics) and metabolomics (e.g., short-chain fatty acids). Saliva and urine will be analyzed for stress-related hormones, metabolomics and specific metabolites of interest. Blood samples will be analyzed for inflammatory cytokines, stress-related hormones, metabolomics, and other potential biomarkers that might be emerging when the sample recruitment is finalized. A subset of participants will undergo a skin punch biopsy to generate a human-derived cell model for investigating causal cellular mechanisms in response to microbial metabolites.

Neurocognitive and neural data will be collected using EEG tasks and computerized cognitive tasks assessing impulsivity and attention.

ELIGIBILITY:
ADHD Group Inclusion Criteria:

1. Be able to give written informed consent
2. Should be stable for 4 weeks on psychopharmacological medication or without medication
3. Should have an established diagnosis of ADHD or ADD as the main mental disorder diagnosis. This will be validated by the ADHD diagnostic criteria after DSM-5, with the DIVA interview.
4. Aged 18-50 years
5. Fluency in English language

Control Group Inclusion Criteria

1. Be able to give written informed consent
2. Should be stable for 4 weeks on any medication for physical health or without medication
3. Should not currently taking psychopharmacological medicine or discontinued psychopharmacological medicine in the past 6 months (due to relapse risk)
4. Should NOT have an established diagnosis or clinical symptoms of ADHD or ADD. This will be validated using with the ASRS-6 (< 4)
5. Should not have a diagnosis of ASD as indicated by self-report.
6. Not have current, or in the past 2 years, symptoms or diagnosis of a depressive disorder, bipolar spectrum disorder, OCD, PTSD, generalised anxiety disorder, severe alcohol or illegal drug dependency, psychotic disorder, anorexia nervosa, and bulimia nervosa
7. Not have current symptoms or diagnosis of a panic disorder or social anxiety disorder that is not currently being treated by a psychotherapist or other mental health care professional
8. Aged 18-50 years
9. Fluency in English language

ADHD and Control Group Exclusion criteria:

1. Current severe depressive (PHQ-9>15), manic or psychotic episode, acute suicidality or suicide attempt in the past 3 months, current severe alcohol and illegal drug dependency as determined by the MINI Psychiatric Interview or clinical diagnosis.
2. Pregnant, breastfeeding, or planning to be pregnant.
3. Habitual fibre intake exceeding 25g/day.
4. Allergy to intervention foods.
5. Allergy to local anaesthesia (only if opting for the skin punch).
6. Taking anticoagulant medication or have coagulation disorder like haemophilia (only if opting for the skin punch).
7. Have a BMI below 18.5 kg/m2.
8. Current diagnosis or symptoms of anorexia nervosa or bulimia nervosa, as determined by clinical diagnosis or on the MINI.
9. Have a significant acute or chronic coexisting illness (cardiovascular, gastrointestinal, endocrinological, immunological, metabolic) or any condition which contraindicates, in the investigator's judgement, entry to the study.
10. Taking antibiotics in the past month (washout period of 1 month is required).
11. Taking medication that the investigator believes would interfere with the objectives of the study, pose a safety risk or confound the interpretation of the study results; to include anti-inflammatory drugs, corticosteroids, laxatives, enemas, anti-coagulants, and over-the counter non-steroidal analgesics. Participants should have a wash-out period of one month.
12. Individuals who, in the opinion of the investigator, are considered to be poor attendees or unlikely for any reason to be able to comply with the trial.
13. Participants receiving treatment involving experimental drugs. Washout period of one month is required.
14. Current prebiotic or probiotic supplement use (a wash-out period of 4 weeks after cessation will allow entry to the study).
15. Previous participation in the Diet Study (APC150)
16. Uncorrected vision.
17. A history of any other condition affecting cognitive function (besides ADHD or ASD for ADHD group participants).

The specific exclusion criteria for electroencephalography (EEG) recording for both the ADHD and Control groups are as follows:

1. Left-handedness,
2. Non-removable medical devices such as pacemakers, hearing aids, cochlear implants, or deep brain stimulators,
3. Hairstyles that prevent access to the scalp, and
4. Skin conditions on the scalp.

Participants who meet these exclusion criteria for the EEG portion of the study will still be included in the overall study but will not undergo EEG recording and will instead complete neurocognitive tasks outside of EEG recording.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Change in ADHD core symptoms | From baseline to 12 weeks
  Change in ADHD core symptoms from baseline to the end of diet (12 weeks) measured by Conner's ADHD rating scale total score (CAARS). The CAARS Total ADHD Symptoms score ranges approximately from 0 to 100, with higher scores indicating greater ADHD symptom severity (worse outcome).

SECONDARY OUTCOMES:
Change in neurocognitive function and mood, and other secondary domains | From baseline to 12 weeks
  Secondary objectives include whether the combined intervention changes neurocognitive function, mood, quality of life, individual goals attainment, changes in sleep, eating behaviour, gastrointestinal symptoms, gut microbial profile, and gut-brain signalling pathways, including immune and inflammatory markers, cortisol, and a broad range of proteins and metabolites.
  Additionally, changes in sub-scales of Conner's ADHD Rating Scale (CAARS) will be assessed as secondary outcome. The sub-scales are: Inattention/Executive Dysfunction (0-30), Hyperactivity (0-13), Impulsivity (0-13), Emotional Dysregulation (0-9), Negative Self-Concept (0-7), with higher scores indicating greater symptom severity (worse outcome).

OTHER OUTCOMES:
Tertiary Outcomes | From baseline to 12 weeks (end of dietary intervention)
  Tertiary outcomes include assessment of the acceptability and feasibility of the combined dietary intervention, validation of a questionnaire assessing the frequency of fermented food intake in adults with and without ADHD, and evaluation of the long-term effects of the intervention on study outcomes at 12 weeks post-intervention.
  Acceptability and feasibility will be assessed using study-specific questionnaire.
  For long-term effects of the intervention, the Conners' Adult ADHD Rating Scales (CAARS) Total ADHD Symptoms will be measured, ranging approximately from 0 to 100, with higher scores indicating greater ADHD symptom severity (worse outcome).

CONTACTS AND LOCATIONS:
Locations (1):
- APC Microbiome Ireland, Cork, Cork, Ireland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Brysbaert M, Stevens M. Power Analysis and Effect Size in Mixed Effects Models: A Tutorial. J Cogn. 2018 Jan 12;1(1):9. doi: 10.5334/joc.10. PMID 31517183
- [Background] Faraone SV, Biederman J, Mick E. The age-dependent decline of attention deficit hyperactivity disorder: a meta-analysis of follow-up studies. Psychol Med. 2006 Feb;36(2):159-65. doi: 10.1017/S003329170500471X. PMID 16420712
- [Background] Konstanti P, Ahrens KF, Neumann RJ, Plichta MM, Schiweck C, Ruf A, Fiebach CJ, Kalisch R, Basten U, Wessa M, Tuescher O, Kollmann B, Lieb K, Arias-Vasquez A, Smidt H, Reif A, Matura S, Belzer C. Impulsivity among healthy adults is associated with diet and fecal microbiota composition. Transl Psychiatry. 2025 Aug 3;15(1):263. doi: 10.1038/s41398-025-03483-4. PMID 40753077
- [Background] Berding K, Cryan JF. Microbiota-targeted interventions for mental health. Curr Opin Psychiatry. 2022 Jan 1;35(1):3-9. doi: 10.1097/YCO.0000000000000758. PMID 34750307
- [Background] Ribera C, Sanchez-Orti JV, Clarke G, Marx W, Morkl S, Balanza-Martinez V. Probiotic, prebiotic, synbiotic and fermented food supplementation in psychiatric disorders: A systematic review of clinical trials. Neurosci Biobehav Rev. 2024 Mar;158:105561. doi: 10.1016/j.neubiorev.2024.105561. Epub 2024 Jan 26. PMID 38280441
- [Background] Bull-Larsen S, Mohajeri MH. The Potential Influence of the Bacterial Microbiome on the Development and Progression of ADHD. Nutrients. 2019 Nov 17;11(11):2805. doi: 10.3390/nu11112805. PMID 31744191